CLINICAL TRIAL: NCT05867732
Title: A Multicenter Observational Cohort of Degenerative Spine Diseases in China
Brief Title: A Multicenter Observational Cohort of Degenerative Spine Diseases in China（DSDC）
Acronym: DSDC
Status: Completed | Type: Observational
Sponsor: Xiamen University (Other)
Responsible Party: Principal Investigator, Wenle Li, Dr., Xiamen University
Other Study IDs: XiamenUDSDC
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Degenerative Spine Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study type: The objectives of this observational study were to understand, analyze, and compare the treatment and prognosis of patients with degenerative spine diseases and to construct a risk warning model and an assisted decision-making system

The main questions it aims to answer are:

* [question 1] to construct a database of patients with degenerative spinal diseases and to study their associated prognosis, complications, and other risks
* [Question 2] Use big data to build a risk early warning model and assisted decision making system The study will not intervene with patients

ELIGIBILITY:
Inclusion criteria:

* patients with degenerative spine disease admitted to the units participating in the study from January 2015 to mid-January 2022;
* complete patient data with no more than 5% missing;

Exclusion Criteria:

* Patients with oncology;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with degenerative spine disease (lumbar disc herniation, lumbar spinal stenosis, lumbar spondylolisthesis, scoliosis deformity, etc.) seen and treated in participating units between January 2015 and January 2022, excluding patients with neoplastic disease
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Collect demographics (Hospital Information System) | 2022.03
  Collect demographics from the HIS system for patients with degenerative spine disease

CONTACTS AND LOCATIONS:
Overall Officials: Wenle Wenle, M.D., Principal Investigator — Xiamen University
Locations (1):
- Wenle Li, Xianmencun, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen N, Zhang Y, Ding Z, Li R, Quan X, Liu X, Zhang Y, Xiang T, Zhang Y, Yin C, Li W. Predicting intraoperative blood loss risk in severe lumbar disc herniation patients undergoing PLIF: a multicenter cohort study using ensemble learning. Int J Surg. 2025 Sep 1;111(9):5904-5913. doi: 10.1097/JS9.0000000000002730. Epub 2025 Jun 19. PMID 40540437
- [Derived] Li W, Zhang Y, Zhou X, Quan X, Chen B, Hou X, Xu Q, He W, Chen L, Liu X, Zhang Y, Xiang T, Li R, Liu Q, Wu SN, Wang K, Liu W, Zheng J, Luan H, Yu X, Chen A, Xu C, Luo T, Hu Z. Ensemble learning-assisted prediction of prolonged hospital length of stay after spine correction surgery: a multi-center cohort study. J Orthop Surg Res. 2024 Feb 2;19(1):112. doi: 10.1186/s13018-024-04576-4. PMID 38308336